CLINICAL TRIAL: NCT07356674
Title: Hemi-tibial Plateau Osteotomy Combined With Arthroscopic Repair for Medial Meniscus Posterior Root Tears in Varus Knees: A Pilot Randomized Controlled Trial
Brief Title: Hemi-tibial Plateau Osteotomy Combined With Arthroscopic Repair for Medial Meniscus Posterior Root Tears in Varus Knees
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eighth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Mengjun Ma, Associate Chief Physician, Department of Orthopaedics, Eighth Affiliated Hospital, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZDBY-IIT-202503-032
Record Dates: First submitted 2025-12-26; First posted 2026-01-21 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Knee Osteoarthristis; Meniscus Injury
Keywords: Hemi-tibial plateau osteotomy; High tibial osteotomy; Medial meniscus posterior root tears; Varus knees

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hemi-tibial plateau osteotomy combined with arthroscopic repair (Experimental)
  Interventions: Procedure: Hemi-tibial plateau osteotomy combined with arthroscopic repair
- High tibial osteotomy combined with arthroscopic repair (Active Comparator)
  Interventions: Procedure: High tibial osteotomy combined with arthroscopic repair

INTERVENTIONS:
Procedure: Hemi-tibial plateau osteotomy combined with arthroscopic repair — The intervention is hemi-tibial plateau osteotomy combined with arthroscopic repair of the medial meniscus posterior root (HTPO combined with arthroscopic repair). After anesthesia and supine positioning, the medial compartment is opened by releasing the distal attachment of the superficial medial collateral ligament. Under fluoroscopic guidance, an L-shaped osteotomy is performed with the horizontal cut approximately 3.0 cm below the tibial plateau, while preserving the articular surface continuity at the hinge area to protect the cartilage and meniscus. A controlled valgus force is then applied to gradually open the osteotomy gap, and the lower-limb alignment is corrected to the preplanned target and confirmed by fluoroscopy. Arthroscopic repair of the medial meniscus posterior root is subsequently performed. The distal attachment of the superficial medial collateral ligament is advanced proximally and fixed below the horizontal osteotomy line, and the osteotomy is stabilized with a
  Arms: Hemi-tibial plateau osteotomy combined with arthroscopic repair
Procedure: High tibial osteotomy combined with arthroscopic repair — The control intervention is high tibial osteotomy combined with arthroscopic repair of the medial meniscus posterior root (HTO combined with arthroscopic repair). After anesthesia and supine positioning, the high tibial osteotomy is performed under fluoroscopic guidance according to the preoperative plan. A controlled valgus force is gradually applied to open the osteotomy gap, and the lower-limb alignment is corrected to the preplanned target and confirmed by fluoroscopy. Arthroscopic evaluation is then performed, followed by arthroscopic repair of the medial meniscus posterior root. The osteotomy site is stabilized with a proximal medial tibial anatomic locking titanium plate, and final fluoroscopic confirmation of alignment and fixation stability is obtained before wound closure.
  Arms: High tibial osteotomy combined with arthroscopic repair

SUMMARY:
This is a single-center clinical trial started by the study team. The goal is to compare two surgeries for people who have a varus knee alignment and a tear at the back attachment of the medial meniscus. Researchers want to learn how the newer bone-cut procedure with arthroscopic meniscus repair compares to the standard bone-cut procedure with arthroscopic meniscus repair. Researchers will also track safety and hospital-related costs.

Main questions the study aims to answer:

* At 12 months after surgery, how does the improvement in knee function compare between the newer-surgery group and the standard-surgery group? The study will evaluate preliminary trends in clinical efficacy using the Lysholm knee function score.
* Do the two groups differ in pain relief, imaging findings, meniscus healing, complications, and hospital stay and preliminary cost-effectiveness? The study plans to enroll about 20 participants at Sun Yat-sen University Eighth Affiliated Hospital (Shenzhen Futian). Participants will be assigned by chance, like drawing lots, in a one-to-one ratio. This is an pilot study with a PROBE (Prospective Randomized Open-label Blinded-Endpoint) design. While participants and surgeons will know which surgery is performed, the research assistant responsible for collecting patient-reported outcomes will be blinded to group allocation to minimize observer bias.

Study groups:

* Experimental group: hemi-tibial plateau osteotomy plus arthroscopic meniscus repair.
* Control group: high tibial osteotomy plus arthroscopic meniscus repair.

Who may join:

* Age 35 to 65 years, with no restriction on sex;
* Diagnosed with a medial meniscus posterior root tear;
* Presence of varus knee deformity;
* Imaging findings support the diagnosis (e.g., knee MRI);
* Failure of conservative treatment: no meaningful improvement after more than 1 month of non-surgical management (e.g., rest, medication, or physical therapy);
* Varus alignment angle less than 10 degrees;
* The deformity is predominantly tibial in origin;
* Knee radiographs do not show the most severe osteoarthritis (Kellgren-Lawrence grade other than IV).

Who cannot join:

* A knee that is chronically "locked," meaning it cannot bend or straighten normally.
* The most severe level of knee arthritis on knee X-ray.
* Severe arthritis in the hip or ankle that could affect knee function testing.
* Inflammatory or infectious conditions that can affect the knee, or abnormal inflammation blood tests that make participation unsafe.
* Knee instability or poorly functioning prior ligament reconstruction, based on the study doctor's judgment.
* Any prior surgery on the target knee, or on other joints of the same-side lower limb.
* Serious heart, liver, or kidney disease, cancer, bleeding disorders, immune deficiency, or severe mental health conditions that make participation unsafe.
* Body mass index of 30 or higher.
* Pregnancy or breastfeeding, or not willing to use birth control during the study.
* Participation in another clinical study within the past 3 months (except registry studies).
* Any other reason the study doctor believes makes participation unsafe or not appropriate.

What participants will do:

* Complete screening and baseline assessments within about 30 days before surgery and sign informed consent.
* Receive the assigned surgery during the hospital stay.
* Return for follow-up visits at 3 months, 6 months, and 12 months after surgery.
* Complete knee function and symptom questionnaires and rate pain at each follow-up visit.
* Have standing knee X-rays and full-length leg X-rays at 3, 6, and 12 months.
* Have an MRI of the operated knee at 3, 6, and 12 months to assess meniscus healing and meniscus extrusion.

Outcomes:

* Primary outcome: change from baseline to 12 months in the Lysholm knee function score.
* Secondary outcomes: changes in the Lysholm score at 3 and 6 months; changes in the WOMAC knee arthritis symptom score at 3, 6, and 12 months; changes in pain rating on a standard pain scale at 3, 6, and 12 months; imaging measures and bone healing on X-rays; meniscus healing and extrusion on MRI; surgery time and blood loss; complications during and after surgery; length of hospital stay and hospital costs; and quality of life utility value from a standard health questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Age 35 to 65 years, with no restriction on sex.
* Clinical features suggestive of a medial meniscus posterior root tear, including at least one of the following symptoms: knee locking, clicking, or medial knee pain; and at least one of the following signs: medial joint line tenderness or a positive McMurray test.
* Varus knee deformity with a varus angle of less than 10 degrees, with the deformity predominantly originating from the tibia (i.e., medial proximal tibial angle less than 87 degrees).
* Knee MRI demonstrates a medial meniscus posterior root tear.
* Knee radiographs show narrowing of the medial joint space, and Kellgren-Lawrence grade less than IV.
* Failure of conservative treatment (e.g., rest, medication, or physical therapy) for more than 1 month.
* Willing to accept randomization and able to understand and sign the informed consent form.
* For participants with bilateral deformity, the more severely deformed side will be selected as the operative (study) side.

Exclusion Criteria:

* Chronic knee locking (e.g., the participant cannot bend or fully straighten the knee).
* Kellgren-Lawrence grade IV knee osteoarthritis.
* Osteoarthritis or other conditions in other joints (e.g., hip or ankle) that may affect assessment of knee function.
* Known inflammatory diseases or other conditions that may affect knee function, including but not limited to: autoimmune diseases (e.g., rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, systemic lupus erythematosus); crystal-induced arthritis (gout, pseudogout); secondary knee osteoarthritis due to trauma or other diseases; active knee joint infection or a history of knee joint infection; reactive arthritis; systemic cartilage disorders; systemic connective tissue diseases; metabolic bone disease; fracture (acute or subacute fracture within 6 months prior to the screening visit); osteonecrosis; or abnormal inflammatory markers (C-reactive protein or high-sensitivity C-reactive protein at least 2 times the upper limit of normal, or erythrocyte sedimentation rate at least 3 times the upper limit of normal), if judged by the investigator to be unsuitable for participation.
* Target-knee instability (including but not limited to post-traumatic or congenital laxity) or inadequate ligament reconstruction, as judged by the investigator.
* Any prior surgery on the target knee or on other joints of the ipsilateral lower limb.
* Serious cardiac disease; hepatic impairment (aspartate aminotransferase or alanine aminotransferase at least 3 times the upper limit of normal, or total serum bilirubin at least 1.5 times the upper limit of normal); renal impairment (serum creatinine at least 1.5 times the upper limit of normal); other musculoskeletal disorders; malignancy; coagulation disorders; immunodeficiency; or psychiatric disorders, if judged by the investigator to be unsuitable for participation.
* Body mass index at least 30 kg/m².
* Pregnant or breastfeeding women, or participants (including men and women) unwilling to use contraception during the study period.
* Participation in another clinical study within 3 months prior to enrollment (excluding registry studies).
* Any other condition that, in the investigator's judgment, makes the participant unsuitable for participation.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Lysholm Knee Score | Baseline (preoperative) and 12 months after surgery
  Lysholm knee score will be assessed preoperatively (baseline) and at 12 months after surgery. The primary endpoint is the change from baseline to 12 months (12-month score minus baseline score). Higher scores indicate better knee function.

SECONDARY OUTCOMES:
Change From Baseline in Lysholm Knee Score (3 and 6 Months) | Baseline (preoperative), 3 months, and 6 months after surgery
  Lysholm knee score will be assessed at baseline (preoperative) and at 3 and 6 months after surgery. The outcome is change from baseline at each time point (score at follow-up minus baseline score). Higher scores indicate better knee function.
Change From Baseline in WOMAC Total Score (3, 6, and 12 Months) | Baseline (preoperative), 3 months, 6 months, and 12 months after surgery
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) total score will be assessed at baseline and at 3, 6, and 12 months after surgery. The outcome is change from baseline at each time point (follow-up minus baseline). WOMAC total score ranges from 0 to 96, with lower scores indicating better symptoms/function.
Change From Baseline in Pain Score (VAS) (3, 6, and 12 Months) | Baseline (preoperative), 3 months, 6 months, and 12 months after surgery
  Pain will be assessed using a 10-cm visual analogue scale (VAS) at baseline and at 3, 6, and 12 months after surgery. The outcome is change from baseline at each time point (follow-up minus baseline). The VAS ranges from 0 (no pain) to 10 (worst pain).
Change in Mechanical Axis Location on Tibial Plateau (%MA) on Full-Length Lower Limb Radiographs | Baseline (preoperative), 3 months, 6 months, and 12 months after surgery
  On bilateral standing full-length lower limb radiographs, the mechanical axis (MA) will be evaluated by the relative location where the mechanical axis crosses the tibial plateau, expressed as a percentage (%MA). The outcome is %MA at each time point and change from baseline.

OTHER OUTCOMES:
Change in EQ-5D-5L Health Utility Value | Baseline (screening/preoperative), 0-7 days after surgery, 3 months, 6 months, and 12 months after surgery
  Health-related quality of life will be assessed using the EQ-5D-5L questionnaire and converted to a health utility value using the China EQ-5D-5L value set. The outcome is the utility value at each time point and change from baseline (follow-up minus baseline).
Quality-Adjusted Life Years (QALYs) Over 12 Months | Baseline to 12 months after surgery
  QALYs will be calculated over the 12-month follow-up period using EQ-5D-5L utility values collected at scheduled visits (area-under-the-curve approach). The outcome is total QALYs accrued from baseline to 12 months.
Change in Kellgren-Lawrence Grade on Knee Radiographs | Baseline (preoperative), 3 months, 6 months, and 12 months after surgery
  Kellgren-Lawrence (K-L) grade will be assessed on knee radiographs at each time point to evaluate radiographic severity of knee osteoarthritis (grades 0-IV). The outcome is K-L grade at each time point.
Bone Healing Grade at the Osteotomy Site (Modified Van Hemert System) | 0-7 days after surgery, 3 months, 6 months, and 12 months after surgery
  Bone healing at the osteotomy site will be graded using a modified Van Hemert system on radiographs. Grades range from 1 to 5, where higher grades indicate more bridging callus and better healing (grade 5 indicates complete bridging). The outcome is healing grade at each time point.
Medial Meniscus Healing Status on MRI | Baseline (preoperative), 3 months, 6 months, and 12 months after surgery
  Medial meniscus posterior root healing will be assessed on MRI and categorized as complete healing, partial healing, or non-healing. Complete healing is defined as continuity of the repaired root seen on all three MRI planes (sagittal, coronal, and axial). Partial healing indicates loss of continuity in any one plane, and non-healing indicates no continuity in any plane. The outcome includes healing category and the proportion of participants in each category at each time point.
Change in Medial Meniscus Extrusion Distance on MRI | Baseline (preoperative), 3 months, 6 months, and 12 months after surgery
  Medial meniscus extrusion will be measured on MRI as the distance between the outer edge of the medial meniscus and the edge of the medial tibial plateau on a standardized reference line. Outcomes include extrusion distance at each time point and change from baseline.
Surgery-Related Outcomes, Complications, and Hospital Resource Use | 0-7 days after surgery; 3 months, 6 months, and 12 months after surgery (complications assessed through 12 months)
  Surgery-related outcomes will include operative time and intraoperative blood loss. Safety outcomes will include intraoperative and postoperative complications (e.g., common peroneal nerve injury, deep vein thrombosis, infection, implant failure, delayed union, or nonunion). Hospital resource use will include length of hospital stay and hospitalization costs. Outcomes will be recorded during the perioperative period and through 12 months after surgery.
Change in Joint Line Convergence Angle (JLCA) on Standing Knee Radiographs | Baseline (preoperative), 3 months, 6 months, and 12 months after surgery
  JLCA will be measured on standing anteroposterior knee radiographs. The outcome is JLCA (degrees) at each time point and change from baseline (follow-up minus baseline).
Change in Medial Joint Space Width (JS) on Standing Knee Radiographs | Baseline (preoperative), 3 months, 6 months, and 12 months after surgery
  Medial joint space width will be measured on standing anteroposterior knee radiographs. The outcome is joint space width (e.g., mm) at each time point and change from baseline (follow-up minus baseline).
Change in Posterior Proximal Tibial Angle (PPTA) on Knee Radiographs | Baseline (preoperative), 3 months, 6 months, and 12 months after surgery
  PPTA will be measured on knee radiographs. The outcome is PPTA (degrees) at each time point and change from baseline (follow-up minus baseline).
Change in Posterior Tibial Slope (PTS) on Lateral Knee Radiographs | Posterior tibial slope will be measured on lateral knee radiographs. The outcome is PTS (degrees) at each time point and change from baseline (follow-up minus baseline).
  Posterior tibial slope will be measured on lateral knee radiographs. The outcome is PTS (degrees) at each time point and change from baseline (follow-up minus baseline).

CONTACTS AND LOCATIONS:
Locations (1):
- The Eighth Affiliated Hospital, Sun Yat-Sen University, Shenzhen, Guangdong, China